CLINICAL TRIAL: NCT07132086
Title: Prospective Observational Study on the Effectiveness of Daridorexant in Chronic Insomnia Using Subjective and Actigraphic Sleep Measures in a Real-World Setting
Brief Title: Prospective Observational Study on the Effectiveness of Daridorexant in Chronic Insomnia in a Real-World Setting
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Enrica Bonanni, Associate Professor of Neurology - Enrica Bonanni, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: 57/2025
Record Dates: First submitted 2025-08-09; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Daridorexant 50 mg orally, once daily at bedtime, administered as monotherapy or add-on therapy for chronic insomnia, in a real-world, observational, prospective clinical setting — Daridorexant 50 mg is administered once daily at bedtime, either as monotherapy or as add-on therapy in patients with chronic insomnia. The intervention is evaluated in a naturalistic, real-world setting over a 3-month observational period. Both subjective (questionnaires, sleep diary) and objective (actigraphy) sleep parameters are collected at baseline, 1 month, and 3 months. Actigraphy is used to assess total sleep time, sleep efficiency, wake after sleep onset, and circadian rhythm parameters. Sleep misperception is calculated as the discrepancy between subjective and objective sleep metrics. The study also explores potential predictors of treatment response such as age, sex, BMI, insomnia duration, and comorbid sleep disorders.
  Other Names: Quviviq 50 mg

SUMMARY:
The primary objectives of this study is to evaluate the real-world effectiveness of daridorexant 50 mg in improving both subjective (self-report) and objective (actigraphic) sleep parameters in patients with chronic insomnia.

The secondary aims of this study are:

* To compare the effectiveness of daridorexant 50 mg with other guideline-recommended therapies for chronic insomnia in improving sleep parameters and sleep health.
* To identify clinical and demographic predictors of response to daridorexant 50 mg, such as age, sex, BMI, duration of insomnia, and treatment regimen (monotherapy vs. add-on).
* To monitor changes over time in the symptoms related to comorbid sleep disorders (e.g., OSA, RLS, circadian rhythm disorders) in patients treated with daridorexant 50 mg.

DETAILED DESCRIPTION:
Insomnia affects approximately 10% of the European population and represents a significant risk factor for multiple chronic conditions, including cardiovascular diseases, depression, and type II diabetes. The latest European Guidelines for the Management of Insomnia have included daridorexant among the first-line pharmacological options for chronic insomnia. Daridorexant is a dual orexin receptor antagonist (DORA) that offers advantages over traditional hypnotics by avoiding common adverse effects such as residual daytime sedation, impaired motor coordination, and the risk of dependence.

Clinical trials have demonstrated that DORAs, including daridorexant, are effective in improving several subjective and objective sleep parameters. However, no studies to date have investigated predictors of treatment response in patients with insomnia receiving daridorexant, despite increasing awareness of the need for personalized pharmacological strategies.

In pivotal trials, daridorexant efficacy was evaluated using both subjective (patient-reported) and objective (polysomnographic) sleep outcomes. While polysomnography (PSG) is the gold standard for objective sleep evaluation, it is poorly suited for long-term, real-world monitoring due to cost, complexity, and reduced ecological validity. In contrast, actigraphy allows for non-invasive, home-based sleep-wake monitoring through wrist movement detection over multiple nights and is widely used in sleep research and clinical settings. However, no studies have employed actigraphy to assess daridorexant's real-world effectiveness, leaving a significant knowledge gap.

Another relevant aspect is the frequent co-occurrence of insomnia with other sleep disorders such as restless legs syndrome (RLS), circadian rhythm sleep-wake disorders, and obstructive sleep apnea (OSA). Evaluating the evolution of symptoms related to these comorbid sleep conditions in patients treated with daridorexant could help clarify whether its use should be expanded or restricted in certain clinical populations.

Study Objectives and Outcome Measures

Primary Objectives:

To evaluate the real-world effectiveness of daridorexant 50 mg in improving both subjective (questionnaire-based) and objective (actigraphy-based) sleep parameters in patients with chronic insomnia.

Secondary Objectives:

To compare the effectiveness of daridorexant 50 mg with other guideline-recommended therapies for chronic insomnia in improving sleep parameters and sleep health.

To identify clinical and demographic predictors of response to daridorexant 50 mg, such as age, sex, BMI, duration of insomnia, and treatment regimen (monotherapy vs. add-on).

To monitor changes over time in the symptoms related to comorbid sleep disorders (e.g., OSA, RLS, circadian rhythm disorders) in patients treated with daridorexant 50 mg.

Primary Endpoint:

This is the first prospective observational study aiming to assess the real-world effectiveness of daridorexant 50 mg in improving both subjective and actigraphic sleep parameters in patients with chronic insomnia. In addition, the study will evaluate possible changes in circadian metrics over time, with the goal of better understanding the impact of daridorexant on patients' sleep-wake rhythm under real-life conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed informed consent form
* Diagnosis of chronic insomnia according to DSM-5 criteria, defined as:

Dissatisfaction with sleep quantity or quality, associated with one or more of the following:

Difficulty initiating sleep

Difficulty maintaining sleep (frequent awakenings or trouble returning to sleep)

Early morning awakenings with inability to return to sleep

The sleep disturbance causes clinically significant distress or impairment in social, occupational, educational, academic, or other important areas of functioning

Sleep difficulties occur despite adequate opportunity and circumstances for sleep

The insomnia is not better explained by or occurring exclusively during other sleep-wake disorders (e.g., narcolepsy, parasomnias, circadian rhythm sleep-wake disorders, breathing-related sleep disorders)

The insomnia is not attributable to the physiological effects of a substance (e.g., drug abuse or medication)

- No contraindications to daridorexant use according to the European Medicines Agency (EMA)

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Withdrawal of informed consent at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with a clinical diagnosis of chronic insomnia according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria, evaluated at the Neurology Clinic of the Azienda Ospedaliero-Universitaria Pisana (AOUP), Italy. Participants will be selected among those who receive a new prescription of daridorexant or another guideline-recommended treatment for insomnia. The population includes individuals with or without comorbid sleep disorders (e.g., RLS, OSA, circadian rhythm disorders). Both treatment-naïve patients and those previously treated with other insomnia therapies may be included, provided they meet inclusion criteria and give informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in total sleep time after 3 months of daridorexant treatment | From baseline (Day 0) to 3 months after treatment initiation
  This outcome assesses the change in both subjective (patient-reported) and objective (actigraphic) total sleep time (TST) from baseline to 3 months after initiating daridorexant 50 mg.
  Primary Outcome Measures:
  * Change in subjective TST [minutes/night]
  * Change in actigraphic TST [minutes/night]
Change in wake after sleep onset after 3 months of daridorexant treatment | From baseline (Day 0) to 3 months after treatment initiation
  This outcome assesses the change in both subjective (patient-reported) and objective (actigraphic) wake after sleep onset (WASO) from baseline to 3 months after initiating daridorexant 50 mg.
  Primary Outcome Measures:
  * Change in subjective WASO [minutes/night]
  * Change in actigraphic WASO [minutes/night]
Change in sleep efficiency after 3 months of daridorexant treatment | From baseline (Day 0) to 3 months after treatment initiation
  This outcome assesses the change in both subjective (patient-reported) and objective (actigraphic) sleep efficiency (SE) from baseline to 3 months after initiating daridorexant 50 mg.
  Primary Outcome Measures:
  * Change in subjective SE. Subjective SE is estimated as the ratio of subjective TST to Time in bed [%]
  * Change in actigraphic SE. Actigraphic SE is estimated as the ratio of actigraphic TST to Time in bed [%]
Change in sleep regularity index after 3 months of daridorexant treatment | From baseline (Day 0) to 3 months after treatment initiation
  This outcome assesses the change in objective (actigraphic) sleep regularity index (SRI) from baseline to 3 months after initiating daridorexant 50 mg.
  Primary Outcome Measure:
  - Change in Sleep Regularity Index (SRI) [%]
Change in self-reported sleep questionnaires after 3 months of daridorexant treatment | From baseline (Day 0) to 3 months after treatment initiation
  This outcome assesses the change in self-reported sleep questionnaires from baseline to 3 months after initiating daridorexant 50 mg.
  Primary Outcome Measures:
  * Change in sleep quality (PSQI score) [range: 0-21]
  * Change in insomnia severity (ISI score) [range: 0-28]
  * Change in daytime functioning and alertness (IDSIQ total score) [range: 0-100]

SECONDARY OUTCOMES:
Change in TST misperception after 3 months of daridorexant treatment | From baseline (Day 0) to 3 months after treatment initiation
  This outcome assesses the change in TST misperception from baseline to 3 months after initiating daridorexant 50 mg.
  TST misperception is calculated as the difference between subjective and actigraphic TST (hours)
Change in SE misperception after 3 months of daridorexant treatment | From baseline (Day 0) to 3 months after treatment initiation
  This outcome assesses the change in SE misperception from baseline to 3 months after initiating daridorexant 50 mg.
  SE misperception is calculated as the difference between subjective and actigraphic SE (%)
Change in WASO misperception after 3 months of daridorexant treatment | From baseline (Day 0) to 3 months after treatment initiation
  This outcome assesses the change in WASO misperception from baseline to 3 months after initiating daridorexant 50 mg.
  WASO misperception is calculated as the difference between subjective and actigraphic WASO (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Enrica Bonanni, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliera Universitaria Pisana, Pisa, Pi, Italy

IPD SHARING:
Plan to Share IPD: No